CLINICAL TRIAL: NCT06090994
Title: A Prospective, Multicenter, Randomized, Parallel Controlled Study Comparing Huaier Granules With Capecitabine Monotherapy for the Prevention of Recurrence and Metastasis After Radical Resection of Stage II Colorectal Cancer
Brief Title: Prevention of Recurrence and Metastasis of Colorectal Cancer by Comparing Huaier With Capecitabine Monotherapy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Sanjun Cai, professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202401
Record Dates: First submitted 2023-10-15; First posted 2023-10-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Cancer
Keywords: Huaier granule; colorectal cancer; capecitabine; recurrence and metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier Granule (Experimental): Oral administration of Huai'er granules, 10g once, 3 times a day, continued until the end of the study, intolerable toxicity, withdrawal from the study for any reason, disease progression or death, whichever occurs first; Or the researcher determines that the subject no longer benefits. It is recommended that Huai'er Granules be used for the first time within 14 days-2 months after surgery. Please refer to the drug instructions for specific usage.
  Interventions: Drug: Huaier granule
- Capecitabine (Active Comparator): Oral administration, 1250mg/m^2, twice a day (2500mg/m^2/d),day 1-14,with one course of treatment every 3 weeks，please refer to the drug instructions for specific usage.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Huaier granule — Oral administration, 10g once, 3 times a day, starting within 14 days-2 months after surgery. Please refer to the medication manual for specific usage.
  Other Names: Z20000109（NMPA Approval Number）
  Arms: Huaier Granule
Drug: Capecitabine — Oral administration, 1250mg/m^2, twice a day (2500mg/m^2/d),day 1-14,with one course of treatment every 3 weeks, for a total of 4-6 courses.
  Arms: Capecitabine

SUMMARY:
This is a prospective, multicenter, randomized, parallel controlled study to evaluate the effectiveness of Huaier Granule in preventing recurrence and metastasis after radical resection of colorectal cancer

DETAILED DESCRIPTION:
It is expected to include 756 patients with colorectal cancer (CRC) who were diagnosed as stage II and underwent radical resection (R0) according to the CSCO colorectal cancer guidelines 2022 and met the criteria for cabetabine monotherapy in the study center from July 2024 to June 2026. The experimental group was treated with Huaier Granule monotherapy, and 378 patients were expected to be included; The control group was treated with capecitabine monotherapy, and 378 cases were expected to be included. Patients in the experimental group began using Huaier granules within 14 days-2 months after surgery. Patients in control group received capecitabine treatment, with one course of treatment every 3 weeks, for a total of 4-6 courses. Patients will be visited every 12 weeks (± 14 days) for the first two years after enrollment, and every 24 weeks (± 14 days) for the third year, until the end of the study, withdrawal from the study for any reason, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, regardless of gender.
* It is diagnosed as colorectal cancer by histopathology, TNM stage Ⅱ.
* Received radical resection of colorectal cancer (R0) within 12 weeks prior to enrollment.
* Not receiving neoadjuvant therapy before surgery, and not receiving any adjuvant therapy after surgery.
* ECOG score 0-2 points.
* According to the CSCO Colorectal Cancer Guidelines 2022, it meets the criteria for receiving monotherapy adjuvant therapy with capecitabine.
* Clear consciousness, language expression or reading ability, able to communicate normally, and cooperate in completing questionnaire assessments.
* Voluntarily join this study and sign an informed consent form.

Exclusion Criteria:

* Low rectal cancer (occurring within 12 centimeters from the anal margin)
* Combining medical history of other malignant tumors.
* Known to be allergic to the components of Huaier granules or avoid or use Huaier granules with caution (only in the experimental group).
* Inability to take orally medication (experimental group, control group with oral medication included in standard treatment plan).
* Pregnant or lactating women or planned pregnancy preparation.
* In the past one month, the subjects have received Huaier granules or traditional Chinese patent medicines and simple preparations with similar efficacy or indications to Huaier granules (such as compound cantharides capsules, cinobufacin capsules, Kangai injection, Pingxiao tablets, please refer to the instruction manual for details).
* Refusal to cooperate with follow-up.
* Other reasons leading to the researcher's belief that it is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival rate (DFS) | start of treatment until 3-year follow-up
  The proportion of surviving patients who did not experience disease recurrence or metastasis within 3 years after R0 surgery.

SECONDARY OUTCOMES:
1-year disease-free survival rate (DFS) | start of treatment until 1-year follow-up
  The proportion of surviving patients who did not experience disease recurrence or metastasis within 1 years after R0 surgery.
2-year disease-free survival rate (DFS) | start of treatment until 2-year follow-up
  The proportion of surviving patients who did not experience disease recurrence or metastasis within 2 years after R0 surgery.
Overall survival (OS) | start of treatment until 3-year follow-up
  The time from randomization and enrollment on the day of the patient to death for any reason.
Quality of Life Score | baseline period and start of treatment until 3-year follow-up
  Evaluation using the EORTC QLQ-C30 (Chinese version) core quality of life scale developed by the European Organization for Cancer Research and Treatment.
The incidence and severity of adverse events (AE) and severe adverse events (SAE) | start of treatment until 3-year follow-up
  The definition and severity grading of AE and SAE refer to the corresponding descriptions in the definition and evaluation section of adverse events, and the incidence rate is defined as the proportion of patients with AE and SAE to the corresponding total population.
The incidence and severity of adverse reactions (ADR), severe adverse reactions (SADR), suspicious and unexpected severe adverse reactions (SUSAR) | start of treatment until 3-year follow-up
  The definition and severity grading of ADR, severe ADR, and SUSAR refer to the corresponding descriptions in the definition and evaluation section of adverse events. The incidence rate is defined as the proportion of patients with ADR, severe ADR, and SUSAR to the corresponding total population.

OTHER OUTCOMES:
Changes in carcinoembryonic antigen (CEA) compared to baseline period (difference) | start of treatment until 3-year follow-up
  The difference in carcinoembryonic antigen levels between the treatment and baseline periods.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjun Cai, PhD, Principal Investigator — Fudan University
Locations (9):
- China (9):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu People's Hospital, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Sanjun Cai, Shanghai, Shanghai Municipality
  - Renji Hospital，Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospita, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No